CLINICAL TRIAL: NCT01206998
Title: Vaginal Progesterone in Patients With Active Preterm Labor
Brief Title: Vaginal Progesterone as a Treatment for Women Active Preterm Labor
Acronym: VagPro
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of support of the drug company for drug and placebo
Sponsor: University of Rochester (Other)
Collaborators: Juniper Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Tulin Ozcan MD, MD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VagPro 27515
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Labor, Premature
Keywords: preterm labor; progesterone; tocolysis; cervical length
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Progesterone; Replens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal progesterone gel (Experimental)
  Interventions: Drug: Vaginal progesterone gel
- Placebo vaginal gel (Placebo Comparator)
  Interventions: Drug: Placebo vaginal gel

INTERVENTIONS:
Drug: Vaginal progesterone gel — Subjects will receive daily vaginal progesterone gel provided by Columbia laboratories (1.125g progesterone gel containing 90mg (8%) progesterone)
  Other Names: Prochieve® 8%/Crinone 8%®
  Arms: Vaginal progesterone gel
Drug: Placebo vaginal gel — Subjects will receive daily placebo vaginal gel, made of an identical bioadhesive delivery system as the active drug
  Other Names: Replens®
  Arms: Placebo vaginal gel

SUMMARY:
The purpose of this study is to compare how well vaginal progesterone works delaying the time to delivery in women with preterm labor compared to placebo. The study will also compare the effect of vaginal progesterone on neonatal outcomes, rate of spontaneous preterm delivery, cervical length and biomarkers of preterm delivery in women diagnosed with and treated with medication to stop preterm labor.

DETAILED DESCRIPTION:
Preterm birth remains a leading cause of perinatal mortality and morbidity. Despite advances in obstetric and pediatric care, the incidence of preterm birth has increased by more than 20% in the last two decades. Approximately 12.8% of births are preterm, however these account for more than 75% of all perinatal morbidity and mortality. Currently prophylactic progesterone administration is the most effective method available for the prevention of recurrent preterm birth. Prior studies have examined the impact of progesterone in women with recurrent preterm birth and cervical shortening. The possible use of progesterone in women experiencing active preterm labor may address the highest risk condition, however, there have not been any clinical trials to date examining this use of vaginal progesterone. Inflammation and decidual hemorrhage are among the proposed mechanisms that appear to be related to preterm labor.We will use a double blinded randomized drug placebo design to study the proposed outcomes in women diagnosed with preterm labor and planned to have standard of care tocolytic therapy. Women will be randomized to daily vaginal progesterone gel or placebo and will be maintained on the drug or placebo until delivery or 36 6/7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Singleton gestation
* Gestational age between 24 0/7 and 33 6/7 weeks of pregnancy by best obstetric estimate
* Preterm labor, defined as more than 6 uterine contractions in 30 minutes associated with cervical change, either shortening and/or dilation by manual exam.
* Management with standard of care tocolytic therapy (nifedipine)
* Planned delivery at Strong Memorial Hospital or Highland Hospital

Exclusion Criteria:

* Cervical dilation more than 4 cm.
* Evidence of rupture of membranes
* Negative fetal fibronectin (if done prior to admission)
* Cervical length greater than 3 cm
* Presence of cervical cerclage
* Major fetal anomaly
* Small for gestational age, i.e., fetuses with estimated fetal weight below the 10th percentile by ultrasound
* Evidence of chorioamnionitis (Temperature >100.4oF with uterine tenderness and maternal or fetal tachycardia or purulent discharge)
* Suspected placental abruption or significant hemorrhage
* Category III fetal heart rate pattern
* Presence of co-existing medical conditions, including maternal diabetes and hypertension and seizure disorder
* Use of any progesterone in current pregnancy within 4 weeks of enrollment
* First dose of standard tocolytic therapy more than 6 hours prior to randomization
* Allergies to progesterone and progesterone gel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Latency to delivery | Time in days from randomization day to day of end of pregnancy

SECONDARY OUTCOMES:
Cervical length | within 24 hours of first tocolytic dose and at first week follow up
Delivery prior to 37, 34 and 32 weeks | after delivery
Number of subsequent hospital admissions for preterm labor | after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tulin Ozcan, MD, Principal Investigator — University of Rochester
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States